CLINICAL TRIAL: NCT06741852
Title: The Diagnostic Yield and Safety of Confocal Laser Endomicroscopy Assisted Endobronchial Ultrasound-guided Mediastinal Cryobiopsy Via a Tunnel for Diagnosing Mediastinal Lymphadenopathy: a Multi-center Randomized Controlled Trial.
Brief Title: Confocal Laser Endomicroscopy Assisted Endobronchial Ultrasound-guided- Transbronchial Mediastinal Cryobiopsy Via a Tunnel for Diagnosing Mediastinal Lymphadenopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China-Japan Friendship Hospital (Other)
Responsible Party: Principal Investigator, Gang Hou, Professor, China-Japan Friendship Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 2024-CLE-LYM
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Mediastinal Lymphadenopathy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participant, investigator, and outcomes accessor was blinded to the intervention.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- nCLE-TBMC via a tunnel (Experimental): Participants will receive nCLE-TBMC to obtain the samples from mediastinal lesions.
  Interventions: Procedure: nCLE assisted endobronchial ultrasound-guided transbronchial mediastinal cryobiopsy via a tunnel
- TBMC via a tunnel (Experimental): Participates will receive TBMC via a tunnel to obtain the samples from mediastinal lesions.
  Interventions: Procedure: Endobronchial ultrasound-guided transbronchial mediastinal cryobiopsy via a tunnel

INTERVENTIONS:
Procedure: nCLE assisted endobronchial ultrasound-guided transbronchial mediastinal cryobiopsy via a tunnel — Patients received 2.5mL of 10% Fluorescite intravenously during nCLE. The CLE probe was preloaded into a puncture dilation catheter and locked into position with 2mm being exposed beyond the tip. puncture dilation catheter. The lymph node was punctured and the needle positioned at its center. The probe was advanced and locked, and the needle was advanced to the contralateral edge of the lymph node. Image acquisition began at the lymph node capsule, and then the subcapsular region, followed by the cortical sinus. When the image showed granuloma or malignant characteristics, the location will be recorded in EBUS, and retract the CLE probe, leaving the sheath of puncture dilation catheter as a tunnel between airway wall and target lymph node. Then, a 1.1-mm cryoprobe was inserted into the target lymph node through this tunnel under the EBUS guidance. The probe was cooled with liquid carbon dioxide for 5-9 seconds. Then retracted with the bronchoscope and the frozen biopsy tissue.
  Arms: nCLE-TBMC via a tunnel
Procedure: Endobronchial ultrasound-guided transbronchial mediastinal cryobiopsy via a tunnel — First a tunnel between airway wall and mediastinal and/or hilar lesion was made by a puncture dilation catheter (BroncTruTM AK-91-55, Broncus Inc. Hangzhou, China). The 1.1mm cryoprobe (Erbe 20402-401, ERBE, Tübingen, Germany) entered the target lymph node through the tunnel under direct monitoring of EBUS, and the distance between the tip of the cryoprobe and the border of target lymph node was measured using EBUS. After confirming that the distance was >5 mm, the probe was cooled with liquid carbon dioxide for 5-9 seconds. Then retracted with the bronchoscope and the frozen biopsy tissue. Samples were retrieved by thawing in saline and then fixed in formalin. The same lymph node was operated for 3 times.
  Arms: TBMC via a tunnel

SUMMARY:
Mediastinal and/or hilar lymphadenopathy (MHL) becoming more and more common in clinical practice with the development of imaging technique. MHL is secondary to various benign and malignant disorders that could be life-threatening conditions due to compression of airways or blood vessels. Accurate and timely diagnosis is important for managing patients with lymphadenopathy. Nowadays, several invasive mediastinal tissue samplings have been designed and development.

For patients with metastatic lymphadenopathy, endobronchial ultrasound (EBUS) guided transbronchial needle aspiration has been recommended as a first-line diagnostic method by several guidelines due to its highly diagnostic sensitivity for non-small cell lung cancer and acceptable safety.However, the relatively limited material retrieved by needle aspiration restricts its diagnostic yield in non-metastatic lymphadenopathy including sarcoidosis, lymphoma, tuberculosis, etc.6,7 It is important to obtain the representative sample which showed the specific pathology for diagnosing patients with non-metastatic lymphadenopathy. Therefore, previous studies attempt to use transbronchial mediastinal cryobiopsy (TBMC) to obtain acquiring samples with sufficient volume suitable for histological and molecular analyses.

Despite several studies have proved that TBMC has a highly diagnostic yield, the heterogeneity of pathologic characteristics in lymph node makes obtaining a representative sample difficult. To overcome the sampling heterogeneity and obtain the possibility of obtaining a representative sample in mediastinal lesions, increasing sampling number had been proved as an effective method in previous studies (5-times TBNA, thrice TBMC). With the increasing sampling number, the potential risk related to the procedure is higher than before.

Needle-based confocal laser endomicroscopy (nCLE) is a laser-based imaging technique that utilizes fluorescence for real-time microscopic imaging at the biopsy needle tip. Compared to EBUS, nCLE enables real-time visualisation of cell shapes, there by acting a real-time microscope. Besides, we had developed a novel procedure which can built a tunnel between airway wall and target lymph node using a puncture dilation catheter and allows various tools to perform procedure, its efficacy and safety had been proved in our published studies.Based on this tunnel, we could perform TBMC under the nCLE guidance. The area with representative pathology of lymph node may be detected by nCLE, and shorten the sampling number. However, it remains unknown which of these techniques is the superior match for needle biopsy.

ELIGIBILITY:
Inclusion Criteria:

* (1) Age ≥18 years old; (2) Patients with at least one mediastinal and/or hilar lymphadenopathy (short-axis ≥1cm that is detected by chest CT or contrast CT; (3) Patients with recently discovered mediastinal lesions, clinical respiratory symptoms of cough, expectoration, thoracalgia, or complicated lung lesions implicated by thoracic image, which indicates the need of biopsy to identify the etiology; (4) Patients who can understand the purpose of the trial, participate voluntarily and sign an informed consent form.

Exclusion Criteria:

* (1) The lesion is a mediastinal cyst or abscess; (2) Combined severe cardiopulmonary diseases, coagulation disorders, poor tolerance to anaesthesia, combined psychiatric disorders or severe neurosis and other relevant contraindications to bronchoscopy; (3) EBUS assessment reveals that the lesion is rich in blood flow or adjacent to a large vessel, etc. Consider biopsy to be high risk and inappropriate for continuation of biopsy; (4) EBUS did not detect lesions in the hilum and/or mediastinum; (5) Those who, in the judgement of the investigator, have poor patient compliance and are unable to complete the study as required due to mental disorders, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield | 14 days post-procedure
  The diagnostic yield was defined as the percentage of biopsy results that matched the final diagnosis.

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Kramer T, Wijsman PC, Kalverda KA, Bonta PI, Annema JT. Advances in bronchoscopic optical coherence tomography and confocal laser endomicroscopy in pulmonary diseases. Curr Opin Pulm Med. 2023 Jan 1;29(1):11-20. doi: 10.1097/MCP.0000000000000929. Epub 2022 Nov 16. PMID 36474462
- [Result] Tournoy TK, Tournoy KG. Digging mediastinal holes with vigour: a word of caution. Eur Respir J. 2021 Dec 31;59(1):2101381. doi: 10.1183/13993003.01381-2021. Print 2022 Jan. No abstract available. PMID 34140295
- [Result] Sun J, Yang H, Teng J, Zhang J, Zhao H, Garfield DH, Han B. Determining factors in diagnosing pulmonary sarcoidosis by endobronchial ultrasound-guided transbronchial needle aspiration. Ann Thorac Surg. 2015 Feb;99(2):441-5. doi: 10.1016/j.athoracsur.2014.09.029. Epub 2014 Dec 12. PMID 25497069
- [Result] Poletti V, Petrarulo S, Piciucchi S, Dubini A, De Grauw AJ, Sultani F, Martinello S, Gonunguntla HK, Ravaglia C. EBUS-guided cryobiopsy in the diagnosis of thoracic disorders. Pulmonology. 2024 Sep-Oct;30(5):459-465. doi: 10.1016/j.pulmoe.2023.11.008. Epub 2024 Jan 5. PMID 38182468
- [Result] Zhang J, Guo JR, Huang ZS, Fu WL, Wu XL, Wu N, Kuebler WM, Herth FJF, Fan Y. Transbronchial mediastinal cryobiopsy in the diagnosis of mediastinal lesions: a randomised trial. Eur Respir J. 2021 Dec 9;58(6):2100055. doi: 10.1183/13993003.00055-2021. Print 2021 Dec. PMID 33958432